CLINICAL TRIAL: NCT02627391
Title: Early Surgery for Patients With Asymptomatic Aortic Stenosis
Acronym: ESTIMATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AOM 140460
Record Dates: First submitted 2015-11-25; First posted 2015-12-10 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Surgery
Keywords: Aortic valve; Stenosis; Surgery
MeSH Terms: conditions — Aortic Valve Stenosis; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early surgery (Experimental): Surgical aortic valve replacement
  Interventions: Other: Early surgical aortic valve replacement
- Delayed surgery according to guidelines (Active Comparator): Surgical aortic valve replacement
  Interventions: Other: Delayed Surgical aortic valve replacement

INTERVENTIONS:
Other: Early surgical aortic valve replacement
  Arms: Early surgery
Other: Delayed Surgical aortic valve replacement
  Arms: Delayed surgery according to guidelines

SUMMARY:
Many cardiologists are convinced that early surgery in asymptomatic aortic stenosis (AS) saves lives. However there is currently no direct evidence for this and most recommendations from the ESC/ EACTS or ACC/ AHA in this field are supported by Level-B or C evidence. Therefore, the investigators designed a randomized controlled trial to demonstrate whether early surgery improves mortality and morbidity of patients with asymptomatic severe AS and low operative risk.

ELIGIBILITY:
Inclusion criteria

* Adult patient, aged between 18 and 80 years (18 ≤ age ≤80)
* Low operative risk, defined as EuroSCORE II ≤ 5%
* No symptom potentially attributable to AS: no dyspnea, angina or syncope during exercise
* No class I indication for surgery
* No symptom/ fall in blood pressure during exercise test
* Severe AS according to current echocardiography criteria: Vmax > 4.0 m/s and/ or MPG > 40 mm Hg); AVA < 1.0 cm2 (not mandatory)
* Preserved LV systolic function: LVEF >50% according to echocardiography ; no LV wall motion abnormality
* Signed informed consent

Exclusion criteria

* Moderate/ high operative risk for aortic valve replacement, defined as EuroSCORE II > 5%
* Class-I indication for AVR (ESC-EACTS 2012, ACC/ AHA 2014) or fall in blood pressure during exercise testing (Class-IIa)
* Other indication for cardiac surgery (CABG, thoracic aorta)
* Positive exercise test including A/ unmasking of symptoms (angina, dyspnea at low workload, dizziness or syncope) during exercise or B/ Fall in systolic blood pressure during exercise below the baseline value.
* Patients unable to perform the exercise ECG
* More than mild AR (>grade 2/4)/ other significant valve disease LVEF ≤ 50%
* Serum creatinine >160 μmol/L
* Serious extra cardiac comorbidity/ life expectancy <2 years
* Patient included in another trial with signed informed consent
* Patient not affiliated to social insurance
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Combination of overall mortality and cardiac morbidity | 1 year after randomization.
  Any adverse cardiac event requiring hospitalization. Adverse cardiac events include: 1/ development of any symptom clearly related to AS (dyspnea, angina, pre-syncope or syncope during exercise); 2/ major adverse cardiac events defined as congestive heart failure or acute coronary syndrome; 3/ death of any cause, including cardiac death.

SECONDARY OUTCOMES:
Each items of the composite criteria, overall and cardiovascular mortality and cardiac morbidity | 1 year after randomization
Number of patients with preserved LV systolic function ( LVEF >50% according to echocardiography ) in each group | assessed at 3 months after surgery
Performance capacities assessed by speckle-tracking imaging (longitudinal function) in each group | assessed at 3 months after surgery
Postoperative Exercise test (Exercise Electrocardiogram) | assessed at 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc MONIN, MD PhD., Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Monin JL, Lancellotti P, Monchi M, Lim P, Weiss E, Pierard L, Gueret P. Risk score for predicting outcome in patients with asymptomatic aortic stenosis. Circulation. 2009 Jul 7;120(1):69-75. doi: 10.1161/CIRCULATIONAHA.108.808857. Epub 2009 Jun 22. PMID 19546391
- [Background] Farre N, Gomez M, Molina L, Cladellas M, Ble M, Roqueta C, Ascoeta MS, Comin-Colet J, Vila J, Bruguera J. Prognostic value of NT-proBNP and an adapted monin score in patients with asymptomatic aortic stenosis. Rev Esp Cardiol (Engl Ed). 2014 Jan;67(1):52-7. doi: 10.1016/j.rec.2013.06.020. Epub 2013 Oct 20. PMID 24774264
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Guyton RA, O'Gara PT, Ruiz CE, Skubas NJ, Sorajja P, Sundt TM 3rd, Thomas JD; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC guideline for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jun 10;63(22):e57-185. doi: 10.1016/j.jacc.2014.02.536. Epub 2014 Mar 3. No abstract available. PMID 24603191
- [Background] Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC); European Association for Cardio-Thoracic Surgery (EACTS); Vahanian A, Alfieri O, Andreotti F, Antunes MJ, Baron-Esquivias G, Baumgartner H, Borger MA, Carrel TP, De Bonis M, Evangelista A, Falk V, Iung B, Lancellotti P, Pierard L, Price S, Schafers HJ, Schuler G, Stepinska J, Swedberg K, Takkenberg J, Von Oppell UO, Windecker S, Zamorano JL, Zembala M. Guidelines on the management of valvular heart disease (version 2012). Eur Heart J. 2012 Oct;33(19):2451-96. doi: 10.1093/eurheartj/ehs109. Epub 2012 Aug 24. No abstract available. PMID 22922415
- [Background] Otto CM, Lind BK, Kitzman DW, Gersh BJ, Siscovick DS. Association of aortic-valve sclerosis with cardiovascular mortality and morbidity in the elderly. N Engl J Med. 1999 Jul 15;341(3):142-7. doi: 10.1056/NEJM199907153410302. PMID 10403851